CLINICAL TRIAL: NCT04217616
Title: Pain Perception, Headache Provocation and Multiomics of People Who Are Unable to Have Headache
Brief Title: Pain Perception of People Who Are Unable to Have Headache
Status: Completed | Type: Observational
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Isa Amalie Olofsson, Medical Doctor, PhD student, Danish Headache Center
Other Study IDs: HR001 Pain
Record Dates: First submitted 2020-01-02; First posted 2020-01-03 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Headache; Pain, Head; Muscle Tenderness; Healthy
Keywords: Headache; Healthy; Muscle Tenderness; quantitative sensory testing; cold pain threshold; heat pain threshold; Total Tenderness Score; Cold Pressor Test; Headache Resistant
MeSH Terms: conditions — Headache; Myalgia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Headache Resistant Participants: Male participants who have never had a headache.
- Non-Resistant Participants: Male participants who have experienced headache. Age matched.

SUMMARY:
Headaches are extremely common illnesses with a combined lifetime prevalence of 90-99% in Europe. Despite this high prevalence, there are persons who have never, in their whole life, encountered a headache.

The aim of the study is to identify factors that protect against headache by studying pain perception, muscle tenderness and pain tolerance in people who never have had a headache (headache resistant) versus non-resistant controls.

The investigators hope to contribute with novelty to the current understanding of headache pathophysiology and development of more efficient treatment of headache.

The investigator examining:

Quantitative sensory testing (cold pain threshold and heat pain threshold), Muscle tenderness (total tenderness score) and cold pressor test (time in the water and pain rating). All tests are performed the same day, by one investigator who are blinded to the grouping of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Headache resistant and non-resistant male participants from the Danish Blood Donor Study.
* Weight: 45 kg to 95 kg

Exclusion Criteria:

* Daily consumption of any medication.
* Consumption of any medication less than 12 hours prior to the study day.
* Headache on the study day or 48 hours prior to the study day.
* Amnestic or clinical signs of hypertension (systolic blood pressure >150 mmHg and/or diastolic blood pressure >100 mmHg) or hypotension (systolic blood pressure <90 mmHg and/or diastolic blood pressure <50 mmHg).
* Any severe cardiovascular disease, including cerebrovascular illness.
* Amnestic or clinical signs of current mental illness.
* Amnestic or clinical signs of current substance or drug abuse.
* Amnestic or clinical signs of any illness the responsible doctor considers relevant for participation in the study.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 Headache resistant and 50 non-resistant male participants from the Danish Blood Donor Study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Quantitative Sensory Test: Cold Pain Threshold | 3 hours
  Difference in Cold Pain Threshold (celcius) between cases and controls.
Quantitative Sensory Test: Heat Pain Threshold | 3 hours.
  Difference in Heat Pain Threshold (celcius) between cases and controls.
Pericranial Muscle Tenderness: Total Tenderness Scores | 3 hours
  Difference in Total Tenderness Score between cases and controls. 8 pericranial muscles are palpated by the investigator and the tenderness is rated by the participant on a scale of 0-3 where 0 is no tenderness and 3 is severe tenderness.

SECONDARY OUTCOMES:
Cold Pressor Test: Pain Tolerance | 3 hours
  Difference in Cold Pressor Test Pain Tolerance (seconds) between cases and controls
Cold Pressor Test: Pain Rating | 3 hours
  Difference in Cold Pressor Test Pain Rating by Verbal Rating Scale (VRS) between cases and controls. The pain is rated by the participant on the Verbal Rating Scale from 0 - 10 where 0 is no pain and 10 is the most severe pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Jes Olesen, Professor, Study Director — Danish Headache Center
Locations (1):
- Danish Headache Center, Glostrup Municipality, Region H, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Olofsson IA, Hvedstrup J, Falkenberg K, Chalmer MA, Schytz HW, Pedersen MB, Ullum H, Pedersen OB, Olesen J, Hansen TF. Pain sensitivity in men who have never experienced a headache: an observer blinded case control study. J Headache Pain. 2021 Nov 8;22(1):134. doi: 10.1186/s10194-021-01345-0. PMID 34749638